CLINICAL TRIAL: NCT03371680
Title: Kinetics of Disaturated-phosphatidylcholine and Specific Surfactant Proteins Turnover, Water Turnover and Total Body Water in Acute Respiratory Distress Syndrome (ARDS) in Intensive Care Unit (ICU) Patients and in Control Patients
Brief Title: Kinetics of Surfactant Proteins, Phosphatidylcholine and Body Water in Intensive Care Unit (ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Città della Speranza, Padova (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1235P
Record Dates: First submitted 2017-10-31; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: ARDS; Sepsis Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection of stable isotopes (Experimental): Injection of 1-13 Carbon Leucine and deuterated water: all patients received a constant intravenous infusion of 1 g 1-13 Carbon Leucine (Cambridge Isotope Laboratories, Andover, MA) dissolved in saline for 24 h. Deuterated water (Cambridge Isotope Laboratories, Andover, MA) was administered as a 25 ml bolus at the study start and then, every 12 hours over the next 36 hours, as intermittent boluses corresponding to 0.0625% of fluid intake, to maintain steady state of deuterium enrichment in body water
  Interventions: Drug: Injection of 1-13 Carbon Leucine and deuterated water

INTERVENTIONS:
Drug: Injection of 1-13 Carbon Leucine and deuterated water — All patients received a constant intravenous infusion of 1 g 1-13 Carbon Leucine (Cambridge Isotope Laboratories, Andover, MA) dissolved in saline for 24 h. Deuterated water (Cambridge Isotope Laboratories, Andover, MA) was administered as a 25 ml bolus at the study start and then, every 12 hours over the next 36 hours, as intermittent boluses corresponding to 0.0625% of fluid intake, to maintain steady state of deuterium enrichment in body water
  Other Names: Isotopes came from Cambridge Isotope Laboratories, MA

SUMMARY:
Analysis of kinetics of phosphatidylcholine and specific surfactant proteins, total body water and water turnover in patients with acute respiratory distress syndrome (ARDS) and in intensive care unit (ICU) patients by using non radioactive isotopes as deuterium and Carbon-13.

DETAILED DESCRIPTION:
Patients with adult respiratory distress syndrome (ARDS) have low concentrations of disaturated-phosphatidylcholine and surfactant protein-B and C in bronchoalveolar lavage fluid and altered fluid metabolism.

Injection of stable isotopes such as 13 Carbon Leucine and deuterated water allows the analysis of disaturated-phosphatidylcholine and surfactant protein-B and C kinetics, total body water and water turnover in patients with ARDS and in human adults with normal lungs (controls).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were:

* adult patients older than 18 years
* expected intensive care unit (ICU) length of stay greater than 120 hours from the onset of acute respiratory failure, defined according to the acute respiratory syndrome (ARDS) Berlin criteria or patients admitted for acute neurological failure defined as Glasgow coma scale < 8.
* All patients with ARDS also had sepsis syndrome or septic shock according to the surviving sepsis campaign criteria at the admission to the ICU, while no patients with acute neurological failure was septic.

At the start of the study, patients with ARDS/sepsis fulfilled also the following criteria:

* start of the study within 72 hours from the onset of the respiratory failure;
* stable hemodynamic conditions, defined as no need of fluid boluses for at least 6 hours before the start of the study;
* serum urea and creatinine within the normal ranges.

Patients with acute neurological failure fulfilled the following inclusion criteria:

* normal chest radiograph;
* arterial partial pressure of oxygen / fraction of inspired oxygen (PaO2/FiO2) >300;
* no evidence of sepsis, according to body temperature, C reactive protein, white cell count and differential count within normal ranges;
* intubation and mechanical ventilation started within 72 h before the beginning of the study.

Exclusion Criteria:

Exclusion criteria for all study subjects were:

* presence of liver failure or renal failure (transaminases > 3 and creatinine > 2 times the normal values),
* burns > 30% of body surface bone marrow or lung transplantation,
* need of fluid boluses to maintain hemodynamic conditions during the study or extracorporeal circulatory support.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Disaturated phosphatidylcholine (DSPC) fractional synthesis rate | 48 hours
  DSPC deuterium incorporation, change from baseline. The following kinetic parameter will be calculated: fractional synthesis rate (expressed as percentage/day)

SECONDARY OUTCOMES:
Disaturated phosphatidylcholine (DSPC) secretion time | 48 hours
  DSPC deuterium incorporation, change from baseline. The following kinetic parameter will be calculated: secretion time (expressed in hours).
Surfactant protein B and Surfactant protein C synthesis rate | 48 hours
  Surfactant protein B and Surfactant protein C 1 -13 Carbon leucine incorporation, change from baseline. The following kinetic parameter will be calculated: fractional synthetic rate (expressed as percentage/day)
Surfactant protein B and Surfactant protein C secretion time | 48 hours
  Surfactant protein B and Surfactant protein C 1 -13 Carbon leucine incorporation, change from baseline. The following kinetic parameter will be calculated: Secretion time (expressed in hours).
Surfactant protein B and Surfactant protein C half life | 48 hours
  Surfactant protein B and Surfactant protein C 1 -13 Carbon leucine incorporation, change from baseline. The following kinetic parameter will be calculated: half life (expressed in hours).
Volume of Total Body water | 10 hours
  Measured by the isotope dilution method using deuterium oxide. Total body water will be expressed in liters

IPD SHARING:
Plan to Share IPD: Undecided